CLINICAL TRIAL: NCT00239629
Title: Differential Effects of Teriparatide and Strontium Ranelate on Bone Remodeling and Formation in Postmenopausal Women With Osteoporosis
Brief Title: Teriparatide and Strontium Ranelate Head-To-Head Comparison Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10080; B3D-EW-GHCX
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide; strontium ranelate

INTERVENTIONS:
Drug: Teriparatide
Drug: Strontium ranelate
Procedure: Transiliac bone biopsy

SUMMARY:
The aim of this study is to directly compare the bone forming effects of 20 microg/day of teriparatide with those of 2 g/day strontium ranelate as measured by the histomorphometric variables and biochemical bone formation markers after 6 months of therapy in postmenopausal women with osteoporosis.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Ambulatory, postmenopausal women aged 45 to 90 years inclusive at the time of entry into the trial, whose last menstrual period or bilateral oophorectomy occurred at least 5 years prior to entry into the trial. Women below the age of 55 years in whom a bilateral oophorectomy cannot clearly be documented must have their postmenopausal status confirmed by a serum FSH level greater or equal to 30 IU/L and serum estradiol level lower or equal to 20 pg/ml or lower or equal to 73 pmol/L.
2. Free of severe or chronically disabling conditions other than osteoporosis.
3. Able to use a pen-type injection delivery system satisfactorily in the opinion of the investigator and willing to be trained on and use the pen-injector on a daily basis.
4. Without language barrier, cooperative, expected to return for all follow-up procedures, and have given informed consent after being informed of the risks, medications, and procedures to be used in the study.
5. Posterior-anterior lumbar spine (L-1 through L-4) BMD and/or femoral neck BMD and/or total hip BMD measurement at least 2.5 standard deviations (SD) below the average bone mass for young women (T-score below or equal to -2.5 standard deviations). The lumbar spine and hip BMD assessment and the determination of the patient's eligibility for entry into the screening phase will be made by the individual investigator. Any lumbar vertebra that cannot be analyzed due to artifacts, severe crush fracture, osteophytes, or other abnormalities, should be excluded from the analysis. A minimum of two lumbar vertebrae in the L-1 through L-4 region must be evaluable by DXA if this is the only anatomical site where the BMD cut-off level less than -2.5 SD is demonstrated. A DXA assessment performed within three months prior to Visit 1 may be acceptable for patient's eligibility.
6. Normal or clinically insignificant abnormal laboratory values (as defined by the investigator) including serum calcium, PTH(1 84), alkaline phosphatase.

   EXCLUSION CRITERIA:
7. History of unresolved skeletal diseases that affect bone metabolism other than postmenopausal osteoporosis including Paget's disease, renal osteodystrophy, osteomalacia, any secondary causes of osteoporosis, hyperparathyroidism (uncorrected), and intestinal malabsorption.
8. In the opinion of the investigator, have any medical or anatomical condition that potentially could put the patient at additional risk of an adverse event due to the biopsy procedure (for example, coagulation abnormality, anticoagulant medication, extreme obesity, etc).
9. Have undergone two previous iliac bone biopsies (one in each iliac crest). Patients with one previous iliac bone biopsy are eligible provided that the new sample is obtained from the contralateral iliac crest.
10. History of malignant neoplasms in the 5 years prior to Visit 1, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated. Patients with carcinoma in situ of the uterine cervix treated definitively more than 1 year prior to entry into the study may be randomized.
11. Increased baseline risk of osteosarcoma; this includes subjects with Paget's disease of the bone, previous primary skeletal malignancy, or skeletal exposure to therapeutic irradiation, i.e. prior external beam or implant radiation therapy. As an elevation of serum skeletal alkaline phosphatase activity may indicate the presence of Paget's disease, an unexplained elevation of this enzyme activity will also be exclusionary.
12. Abnormal thyroid function not corrected by therapy. Normal thyroid function may be documented by a normal TSH during the screening phase or a combination of clinical and biochemical parameters which, in the judgment of the investigator and the Lilly Clinical Research Physician, sufficiently establishes the presence of normal thyroid function.
13. Active liver disease or clinical jaundice.
14. Significantly impaired renal function as defined by either of the following criteria:

    * Serum creatinine that, in the opinion of the investigator, indicates significant renal impairment.
    * Measured or calculated endogenous creatinine clearance less than 30 mL/min using the following Cockcroft Gault formula for creatinine clearance (ClCr) for women:

    ClCr (mL/minute) = [[(140-age) x weight (kg)]x0.85] / [72 x serum Cr (mg/dL)]
15. Current or past treatment with any bisphosphonate, parathyroid hormone or its analogs, androgens or other anabolic steroids or therapeutic doses of fluorides at any time prior to Visit 2.

    Past treatment (more than 12 months before Visit 2) with a selective estrogen receptor modulator (SERM), nasal or injectable calcitonin, oral, transdermal, or injectable estrogens, progestins, estrogen analogs, estrogen agonists, estrogen antagonists or tibolone is allowed. Previous or current use of fluoridated water or topical dental fluoride treatments are permitted.
16. Treatment with Vitamin D greater than 50,000 IU/week, or with any dose of calcitriol or Vitamin D analogs or agonists in the 6 months prior to Visit 2.
17. Treatment with systemic corticosteroids in the last month prior to Visit 2 or for more than 14 days in the 1 year prior to Visit 2. Ophthalmic, otic, topical, orally inhaled, nasally inhaled, or intra-articular corticosteroid therapy may be used without these restrictions. However, orally inhaled or nasally inhaled corticosteroids in doses greater than 840 micrograms/day beclomethasone dipropionate or equivalent for more than 14 days in the last year prior to randomization will be disqualifying.

Ages: 45 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73
Dates: Start 2005-09; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy measure is the mineralization surface (MS%BS) evaluated in double tetracycline stained bone biopsies.

SECONDARY OUTCOMES:
Other routine histomorphometric parameters, measured at visits 2, 3, 4, and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague, Czechia
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vogelsang
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kifissia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa, Israel
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara, Mexico
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com